CLINICAL TRIAL: NCT06402240
Title: Feasibility, Acceptability, and Potential Efficacy of an Adjunct Digital Health Solution to Standard Dialectical Behavior Therapy
Brief Title: The Pocket Skills Adjunct Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Windsor (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Alexander Daros, Assistant Professor, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 166/2023
Record Dates: First submitted 2024-01-05; First posted 2024-05-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Substance Use Disorders; Alcohol Use Disorder; Depression; Anxiety
Keywords: dialectical behavior therapy; substance use disorders; internet-delivered; adjunct intervention; alcohol use disorder
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Depression; Anxiety Disorders | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Pragmatic single-arm clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adjunct Intervention (Experimental): The intervention is called Pocket Skills 2.0, which is a web-based dialectical behavior therapy skills training (DBT-ST) intervention. The content and material is based on the most recent Linehan (2014) DBT-ST manual. Pocket Skills 2.0 incorporates brief lessons using videos featuring Dr. Linehan herself, exercises involving interaction with the chatbot which allow for text input and selection of responses, and the ability to gain points and unlock additional content which increases user engagement. Pocket Skills is currently the only comprehensive and not-for-profit DBT-ST app available where the effectiveness has been evaluated in at least three research trials.
  Interventions: Behavioral: Dialectical Behavior Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — Dialectical behavior therapy (DBT) in its fully adherent form is a comprehensive intervention involving individual, group, and phone coaching sessions that addresses complex psychological conditions including suicidality, personality disorders, and post-traumatic stress disorder. Evidence for briefer formats incorporating the group skills training format have been successful for many types of conditions, which includes alcohol and substance use disorders. DBT skills training (DBT-ST) involves structured lessons for learning skills in 5 areas: mindfulness, emotion regulation, distress tolerance, interpersonal effectiveness, and addiction. The current intervention is an internet-delivered version of DBT-ST which aims to teach people the same 5 areas of skills in an online environment with a chatbot and interactive format.

SUMMARY:
This study aims to provide access to an adjunct intervention alongside standard group DBT services to examine feasibility, acceptability, and potential added efficacy of the adjunct. The adjunct intervention is an online tool based on DBT skills training and was already evaluated as a self-guided intervention. Participants will complete a baseline session and be given immediate access to the adjunct intervention. Participants will be followed for 12 weeks and complete assessments every 4 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the potential benefits of an optional add-on tool (i.e., an additional tool participants can use at the same time) alongside standard dialectical behavior therapy (DBT) group treatment (i.e., skills training). The adjunct tool is an online website that participants can use on any device connected to the internet and is also based on DBT.

The proposed study will be a single-arm pragmatic clinical trial aiming to recruit 30 participants over the course of 12 months. Participation in this research study includes a telephone screening visit, informed consent, and baseline assessment visit (conducted via video conferencing). Following the baseline assessment there will be three follow-up assessments completed remotely at weeks 4, 8, and 12.

The adjunct intervention is Pocket Skills 2.0, a skills training app based on dialectical behavior therapy. Participants receive access to this tool in conjunction with their start of standard dialectical behavior therapy. A member of the research team will help participants sign-in for the first time. The tool can be used in any internet browser on any device connected to the internet (e.g., computer, smartphone, tablet). Participants are expected to use the app at least twice a week.

At baseline, a brief interview is completed, along with some questionnaires online. Participants are also asked about the treatment they recently started/plan to start. The interview (40-60 minutes) will involve questions about background, treatment history, and current and past psychological symptoms, and history of substance use. The questionnaires ask a range of questions related to mood, and difficulties with functioning, among other questions. These questions should only take about 15-20 minutes to answer and should be completed within 24 hours.

Participants receive requests to complete additional questionnaires online on three additional occasions (week 4, 8, and 12). Links to the questionnaire package will be sent via email (or text) and they will involve questions about well-being as well as a chance to provide open-ended feedback on the app itself. These surveys will take roughly 15-20 minutes. After 12 weeks, participants are reimbursed for their time.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 to 70
2. Fluency in English.
3. Understanding and willingness to comply with study requirements / capable of providing autonomous informed consent.
4. Smartphone or tablet capable of downloading and running the web application, or a computer with access to the internet.
5. Past year alcohol or substance use disorder
6. Use of alcohol or substance in the past month.
7. Starting DBT or has started DBT within the last 15 days.
8. Reports at least "contemplation" levels (score of 4+) of change with respect to substance use problems.

Exclusion Criteria:

1. Any known practical factors that would preclude participation (e.g., extended absences) in the study.
2. Acute psychiatric (e.g., psychosis, mania) or medical condition (including acute intoxication or withdrawal requiring medical attention) that precludes participation in this study.
3. Participation in another treatment/intervention study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Severity of Dependence Scale | 30 days
  Level of dependence on most problematic substance over past 30 days. Minimum score: 0, maximum score 15. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (Depression Subscale; PHQ-9) | 14 days
  Level of depressive symptoms over the past 14 days. Minimum score: 0, maximum score 27. Higher scores mean worse outcome.
Generalized Anxiety Disorder-7 (GAD-7) Scale | 14 days
  Level of generalized anxiety symptoms over the past 14 days. Minimum score: 0, maximum score 21. Higher scores mean worse outcome.
Difficulties in Emotion Regulation Scale, Short Form (DERS-SF; Kaufmann et al., 2015) | 30 days
  Level of emotion dysregulation or the difficulty in changing unwanted emotions effectively in the past month. Minimum score: 18, maximum score 90. Higher scores mean worse outcome.
WHO Disability Assessment Schedule Short Form (WHODAS 2.0) | 30 days
  Level of functional disability in the past month. Minimum score: 0, maximum score 48. Higher scores mean worse outcome.
Mindful Attention and Awareness Scale (MAAS) | 30 days
  Measure of core mindfulness skills around awareness and acceptance, over the past month. Minimum score: 0, maximum score 6 (mean score on 15 items). Higher scores indicate more positive outcome (e.g., more mindful awareness).
Suicidal Behaviors Questionnaire, Revised (SBQ-R; Osman et al., 2001) | 30 days
  Measure of suicidal ideation and behaviors over the past month. Minimum score: 3, maximum score: 18. Higher scores indicate worse outcome.
Risky, Impulsive, and Self-Destructive Questionnaire (RISQ) | 30 days
  Measure of risky and impulsive behavior, past month. Only subscales pertaining to sexual behavior and general reckless behavior will be used. Minimum score: 0, Maximum score: 40. Higher scores indicate worse outcome (e.g., more impulsive and/or risky behaviors)
NIDA Assist | 30 days
  Assesses the frequency of non-alcohol substance use over the past month. Minimum score per item: never used substance; maximum score per item: used substance daily or almost daily. Higher scores indicate worse outcome (e.g., more substance use).
Daily Drinking Questionnaire (DDQ) | 30 days
  Assesses the frequency and quantity of alcohol use and binge drinking episodes over the past month. Minimum score: no alcoholic drinks on specific day; Maximum score: 15+ drinks on a specific day. Higher scores indicate worse outcome (E.g., more alcoholic drinks consumed).
Dialectical Behavioral Therapy Ways of Coping Checklist | 30 days
  Assesses the frequency and intensity of using DBT skills in the past month. Investigators will use the DBT skills subscale only with an average score of 38 items presented. Higher scores indicate greater use of DBT skills.

OTHER OUTCOMES:
Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000) | Baseline only
  Measure of treatment credibility and expectancy for interventions. Minimum score: 4; Maximum score: 56; Higher scores mean participants perceive the intervention to provide expected benefits and/or improvements.
Treatment Acceptability Questionnaire (TAQ; Hunsley, 1992) | 30 days
  Whether or not the treatment is seen as acceptable and helpful with respect to current symptoms/problems. Minimum score: 6, maximum score: 42. Higher scores indicate better treatment acceptability and positive perceptions of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data can be shared upon request. An open-access database will be created to store data within 2 years of study completion.